CLINICAL TRIAL: NCT06836830
Title: Peri-Arrest Ventilation With Positive End-Expiratory-Pressure vs. Zero End-Expiratory-Pressure in Out-of-Hospital-Cardiac-Arrest
Brief Title: PEEP vs. ZEEP in Out-of-Hospital-Cardiac-Arrest
Acronym: PerAVent
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muehlenkreiskliniken, MKK (Other)
Responsible Party: Principal Investigator, Gerrit Jansen, Principal Investigator, Muehlenkreiskliniken, MKK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-1148
Record Dates: First submitted 2025-01-21; First posted 2025-02-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Ventilation Therapy; PEEP, Occult; CPR; Cardiac Arrest (CA)
Keywords: Cardiac Arrest; Positive End-Expiratory Pressure; Zero End-Expiratory Pressure; Ventilation; Randomized Controlled Trial; Emergency Medicine; Resuscitation; CPR
MeSH Terms: conditions — Positive-Pressure Respiration, Intrinsic; Heart Arrest; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEEP (Experimental): PEEP Group (Intervention Group): Patients will receive mechanical ventilation with end-expiratory-pressure set at 5 mbar (PEEP).
  Interventions: Procedure: PEEP 5 mbar
- ZEEP (Experimental): ZEEP Group (Control Group): Patients will receive mechanical ventilation with end-expiratory-pressure set at 0 mbar (ZEEP).
  Interventions: Procedure: ZEEP 0 mbar

INTERVENTIONS:
Procedure: PEEP 5 mbar — Positiv-End-Expiratory Pressure
  Arms: PEEP
Procedure: ZEEP 0 mbar — Zero-End-Expiratory Pressure
  Arms: ZEEP

SUMMARY:
Out-of-hospital cardiac arrest (OHCA) remains a major cause of mortality, with low survival probabilities to hospital discharge. Despite the frequent use of airway management and mechanical ventilation during resuscitation, there is limited evidence regarding the optimal ventilation strategy to improve oxygen delivery and patient outcomes. The present study aims to investigate the effects of positive-end-expiratory-pressure (PEEP) set at 5 mbar compared to zero-end-expiratory-pressure (ZEEP) on the return of spontaneous-circulation (ROSC) in adult patients with OHCA.

DETAILED DESCRIPTION:
This is a prospective, multicenter, cluster-randomized controlled trial conducted across emergency medical services (EMS) in the regions of Guetersloh, Minden-Luebbecke and Osnabrueck. Adult patients (>= 18 years) with OHCA who are undergoing mechanical ventilation through an airway device will be enrolled. The clusters (regional district) will be randomized into two groups: one group will receive ventilation with PEEP set at 5 mbar (intervention group), while the other group will receive ventilation with ZEEP (control group). The study's primary endpoint is the rate of ROSC. Secondary endpoints include rate of re-arrest, death during pre-hospital care phase, hospital admission during ongoing resuscitation, hospital admission with spontaneous circulation, peripheral oxygen saturation and end tidal CO2 at hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years
* non-traumatic OHCA
* mechanical ventilation via airway device

Exclusion Criteria:

* Patients < 18 years,
* traumatic cause of OHCA,
* no cardiac arrest, withholding of resuscitation (e.g. Do-Not-Resuscitate orders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The return of spontaneous circulation (ROSC) | During or after resuscitation
  The primary outcome is the ROSC, defined according to the Utstein template by the presence of a palpable pulse during or after resuscitation. This will be measured as a binary outcome (palpable pulse, yes or no).

SECONDARY OUTCOMES:
Re-Arrest-Rate | Upon hospital admission
  Any need for chest compressions after ROSC (yes vs. no)
Death during pre-hospital care phase | Upon hospital admission
  Any death during pre-hospital care phase (yes vs. no)
Hospital admission during ongoing resuscitation | at hospital admission
  Need for chest-compressions at hospital admission (yes vs. no)
Hospital admission with spontaneous circulation | at hospital admission
  Hospital admission with spontaneous circulation without need for chest compressions (yes vs. no)
SpO2 at hospital admission | at hospital admission
  SpO2 at hospital admission (%)
FiO2 at hospital admission | at hospital admission
  FiO2 at hospital admission (%)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Emergency Medical Services, Gütersloh, North Rhine-Westphalia
  - JWK Minden, Minden, North Rhine-Westphalia
  - Emergency Medical Services, Osnabrück

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vaseekaran M, Vollmer T, Kolaparambil Varghese LJ, Zeichen C, Hinkelbein J, Abels R, Strickmann B, Deicke M, Grannemann JJ, Grunzig R, Hoyer A, Persson J, Tiesmeier J, Veit G, Jansen G. Peri-arrest ventilation with positive end-expiratory-pressure vs. zero end-expiratory-pressure in out-of-hospital-cardiac-arrest (PerAVent)-a prospective, cluster-randomized multicenter trial. Trials. 2026 Jan 21;27(1):69. doi: 10.1186/s13063-025-09292-w. PMID 41566395